CLINICAL TRIAL: NCT01585285
Title: Composite Arterial and Venous Grafting Strategy Versus Conventional Coronary Artery Bypass Grafting for the Anterolateral Territory: a Prospective Randomized Clinical Trial
Brief Title: Coronary Artery Bypass Grafting Strategies for the Anterolateral Territory: a Prospective Randomized Clinical Trial
Acronym: AMI-PONT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUM-11-233
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass grafting; Left internal mammary artery; Composite grafting; Multislice Spiral Computed Tomography Scanner; Graft patency assessment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIMA to SVG Bridge (Experimental): Patients will receive composite coronary artery bypass grafting (CABG) with left internal mammary artery (LIMA) and saphenous vein graft (SVG) Bridge for the anterolateral targets
  Interventions: Procedure: LIMA to SVG Bridge Technique
- Conventional CABG (Active Comparator): Patients will receive conventional coronary artery bypass grafting (CABG) with left internal mammary artery (LIMA) graft to the left anterior descending (LAD) and separate sequential aorto-coronary saphenous vein grafts (SVG) to the others anterolateral targets
  Interventions: Procedure: Conventional CABG

INTERVENTIONS:
Procedure: LIMA to SVG Bridge Technique — This surgical design use a composite-sequential venous graft to distribute left internal mammary artery (LIMA) inflow directly to the left anterior descending (LAD), but also to the other branches of the anterolateral territory thereby promoting a higher flow through the LIMA pedicle. It is constructed using a short saphenous vein graft (SVG) bridge interposed between the LAD and one (or more) other anterolateral targets, with the LIMA grafted on the hood of the SVG just above the LAD anastomosis.
  Arms: LIMA to SVG Bridge
Procedure: Conventional CABG — Conventional coronary artery bypass grafting (CABG) strategy with left internal mammary artery (LIMA) graft to the left anterior descending (LAD) and separate sequential aorto-coronary saphenous vein grafts (SVG) to the others anterolateral targets
  Arms: Conventional CABG

SUMMARY:
The purpose of the AMI-PONT trial is to assess whether the results in term of graft patency with a novel coronary artery bypass (CABG) strategy, including a saphenous vein bridge to distribute the arterial flow of the left anterior mammary artery (LIMA) to all the anterolateral territory, are not inferior than a conventional CABG strategy combining separated LIMA graft to left anterior descending coronary and vein graft for other target vessels of the anterolateral territory.

DETAILED DESCRIPTION:
Purpose: This novel surgical design use a composite-sequential venous graft to distribute left anterior mammary artery (LIMA) inflow directly to the left anterior descending coronary (LAD), but also to the other branches of the anterolateral territory thereby promoting a higher flow through the LIMA pedicle. It is constructed using a short saphenous vein graft (SVG) bridge (LSVB) interposed between the LAD and one (or more) other anterolateral targets, with the LIMA grafted on the hood of the SVG just above the LAD anastomosis.

Objectives. The main objective of the prospective randomized clinical trial AMI-PONT is to assess whether a CABG strategy including a LSVB to distribute the LIMA outflow provides non-inferior patency rates compared to conventional CABG surgery with separated LIMA graft to LAD and SVG to other anterolateral targets.

Methods. Two hundred adult patients undergoing primary isolated CABG, requiring grafting of LAD and at least one other anterolateral target, will be randomized 1:1 in two treatment arms: 1) CABG strategy with LSVB; and 2) conventional CABG strategy with LIMA graft to the LAD and separate aorto-coronary SVG to other anterolateral targets. Patients will be assessed clinically at 30 days, 6 months, one, five and ten years. They will undergo graft patency assessment at one and five years using Multi-Slice Computed Tomography. All patients will undergo CABG using cardiopulmonary bypass (CPB). Patients will be excluded if they have a contraindication to CPB or MSCT graft assessment.

ELIGIBILITY:
Inclusion Criteria: Patients who undergo coronary artery bypass grafting (CABG) surgery (for single, double or triple vessel disease) will be eligible if they:

1. require isolated CABG with median sternotomy on at least one left anterior descending (LAD) site and another anterolateral target;
2. provide written informed consent;
3. are more than 21 years of age.

Exclusion Criteria: A patient will be excluded from the study if he/she does not fulfill the inclusion criteria, the patient or the treating physician refuse the study or if any of the following are observed:

1. concomitant cardiac procedure associated with CABG including valve surgery and ascending aorta surgery;
2. contra-indications to cardiopulmonary bypass (calcified aorta);
3. unusable left internal mammary artery (LIMA) such as uncorrected subclavian artery stenosis, anterior chest trauma, radiation or injury during harvesting precluding the use of the LIMA;
4. concomitant life-threatening disease likely to limit life expectancy to less than 2 years;
5. emergency CABG surgery (immediate revascularization for hemodynamic instability precluding patient consent);
6. prior CABG;
7. severe congestive heart failure with left ventricular ejection fraction less than 30%.

   Other exclusion criteria precluding MSCT include:
8. moderate to severe renal impairment (estimated glomerular filtration rate, eGFR <50 mL/min/1.73 m2);
9. chronic atrial fibrillation (which can preclude ECG-gating during MSCT);
10. history of severe hypersensitivity to iodinated contrast agents;
11. known or suspected for pheochromocytoma;
12. pregnant/lactating female.

    Furthermore, patients may be excluded at the time of MSCT if they are:
13. in persistent rapid (>100/min) atrial fibrillation or any other cardiac rhythm that precludes reliable ECG triggering;
14. severe congestive heart failure, New York Heart Association (NYHA) Class IV, despite coronary revascularization and maximal medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-07; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Anterolateral territory graft patency index | 1 year
  Proportion of patent (non-occluded) distal anastomoses out of the total number of distal anastomoses for anterolateral distribution including the LAD and the other anterolateral territory coronary target assessed by multi-slice computed tomography angiography for all patients

SECONDARY OUTCOMES:
Assessment of grafts patency taken separately | 1 and 5 years
  LIMA to LAD graft patency will be specifically assessed in both groups. Since the grafting strategy provides direct perfusion of the LAD by anastomosing on the hood of the SVG anastomosis to the LAD, we do not expect to see a difference between groups for the expected superior LIMA-LAD patency
Composite clinical outcome | 30 days, 1, 5 and 10 years
  Occurrence of the composite outcome of total mortality, nonfatal myocardial infarction, or target vessel revascularization (i.e. redo CABG surgery or percutaneous coronary intervention). Each clinical outcome will also be assessed separately.
Cardiovascular mortality | 30 days, 1, 5 and 10 years
  Cardiovascular (CV) mortality: all deaths after the first 30 days are considered CV deaths unless a specific non-cardiovascular cause is evident and considered to be the cause of death (e.g. malignancy). Furthermore, patients who die during the index hospitalization but after the initial 30 days period (i.e. long ICU stay with sepsis) will be considered as CV deaths.
Recurrence of angina | 30 days, 1, 5 and 10 years
  Recurrence of angina: new onset of typical chest angina with documented ischemia by stress testing (ECG, echocardiography, or nuclear) or persistence of CCS grade ≥2 angina after surgery.
Anterolateral territory graft patency index | 5 years
  Proportion of patent (non-occluded) distal anastomoses out of the total number of distal anastomoses for anterolateral distribution including the LAD and the other anterolateral territory coronary target assessed by multi-slice computed tomography angiography for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Mathieu Stevens, MD, PhD (c), Principal Investigator — Centre Hospitalier de l'Universite de Montreal (CHUM)
Locations (1):
- Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Manuscripts, Abstracts, Presentations
Time Frame: The study was presented at the EACTS meeting in Milan Oct 2022
Access Criteria: Access to Journal

REFERENCES:
- [Background] Drouin A, Noiseux N, Chartrand-Lefebvre C, Soulez G, Mansour S, Tremblay JA, Basile F, Prieto I, Stevens LM. Composite versus conventional coronary artery bypass grafting strategy for the anterolateral territory: study protocol for a randomized controlled trial. Trials. 2013 Aug 26;14:270. doi: 10.1186/1745-6215-14-270. PMID 23971858
- [Background] Tremblay JA, Stevens LM, Chartrand-Lefebvre C, Chandonnet M, Mansour S, Soulez G, Prieto I, Basile F, Noiseux N. A novel composite coronary bypass graft strategy: the saphenous vein bridge--a pilot study. Eur J Cardiothorac Surg. 2013 Oct;44(4):e302-7. doi: 10.1093/ejcts/ezt388. Epub 2013 Jul 31. PMID 23904134
- [Derived] Stevens LM, Chartrand-Lefebvre C, Mansour S, Beland V, Soulez G, Forcillo J, Basile F, Prieto I, Noiseux N. Anterolateral territory coronary artery bypass grafting strategies: a non-inferiority randomized clinical trial: the AMI-PONT trial. Eur J Cardiothorac Surg. 2023 Apr 3;63(4):ezad060. doi: 10.1093/ejcts/ezad060. PMID 36805638